CLINICAL TRIAL: NCT04399382
Title: A Clinical Study Using Damage-associated Molecular Pattern and Apparent Diffusion Coefficient to Evaluate the Efficacy of Biologics for Treating Spondyloarthritis
Brief Title: A Clinical Study to Evaluate the Efficacy of Biologics in SpA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HKUSZH201902013
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Spondyloarthritis (SpA)
Keywords: MRI; Apparent Diffusion Coefficient; Biomarker; Damage-Associated Molecular Pattern; Chinese
MeSH Terms: conditions — Spondylarthritis | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-radiographic group: Participants with non-radiographic axial SpA
  Interventions: Drug: Biologics
- Radiographic group: Participants with radiographic axial SpA (a.k.a. ankylosing spondylitis)
  Interventions: Drug: Biologics

INTERVENTIONS:
Drug: Biologics — The exposure of interest in this observational study is the biological therapy of Tumor Necrosis Factor (TNF) inhibitor, specifically etanercept biosmilar/ infliximab/ adalimumab/ golimumab.

SUMMARY:
Spondyloarthritis (SpA) is one of the potentially debilitating inflammatory diseases that affect the whole body, primarily burdening the sacroiliac joints and the spine. It mostly affects young and middle aged adults. SpA can be classified to non-radiographic axial SpA (nr-axSpA) and radiographic axSpA (r-axSpA). The latter is ankylosing spondylitis (AS). The key to its early treatment is the radiological detection and management of sacroiliitis. To date, biologics is the most powerful anti-inflammatory drug. Recent research has shown that diffusion-weighted imaging (DWI) outperforms the sequence recommended by the Guidelines in diagnosing inflammation and assessing disease activity. Preliminary research conducted by our team has also demonstrated that apparent diffusion coefficient (ADC) is a valuable imaging biomarker. However, to date, no serum maker of comparable effectiveness has been identified. Damage-Associated Molecular Pattern (DAMP), including S100A8 and S100A9, high mobility group protein B1 (HMGB1) and Tenascin-C (TNC), may play a role in inflammation by regulating the TLR4/MyD88/NF-κB signaling pathways. The present study will enroll 20 patients with nr-axSpA and 20 patients with AS. It will utilize serum DAMP and ADC to assess disease activity before and after treatment as well as the change in and correlations of treatment outcomes, in order to identify objective and quantifiable serum and imaging markers that are beneficial in clinical applications. ADC is the primary outcome. The main hypothesis is that disease activity as measured by ADC will be reduced after 1 year of treatment from baseline as compared to before treatment at baseline. Study findings will indicate the utility of ADC as an objective indicator of disease activity for guiding therapeutic approaches and improving dosage adjustment in clinical applications.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with non-radiographic or radiographic axial SpA

Exclusion Criteria:

* Unable to provide written consent
* Unable to undergo MRI examination
* Pregnancy
* Unable to read and/or write Chinese

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with axial SpA who attend the rheumatology clinic of The University of Hong Kong-Shenzhen Hospital will be screened consecutively by the PI, her trained nurses, and/or research assistants for eligibility. Eligible patients will be recruited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Apparent Diffusion Coefficient | 1 year
  Apparent Diffusion Coefficient (ADC)

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Xian, Shenzhen, Guangdong / 广东, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lecouvet FE, Vander Maren N, Collette L, Michoux N, Triqueneaux P, Stoenoiu M, Houssiau F, Malghem J, Denis ML, Larbi A, Nzeusseu Toukap A. Whole body MRI in spondyloarthritis (SpA): Preliminary results suggest that DWI outperforms STIR for lesion detection. Eur Radiol. 2018 Oct;28(10):4163-4173. doi: 10.1007/s00330-018-5377-3. Epub 2018 Apr 17. PMID 29666994
- [Background] Wang F, Chu C, Zhu L, Zhao C, Wei Y, Chen W, He J, Sun L, Zhou Z. Whole-lesion ADC histogram analysis and the spondyloarthritis research consortium of canada (SPARCC) MRI index in evaluating the disease activity of ankylosing spondylitis. J Magn Reson Imaging. 2019 Jul;50(1):114-126. doi: 10.1002/jmri.26568. Epub 2018 Dec 16. PMID 30556229
- [Background] Bradbury LA, Hollis KA, Gautier B, Shankaranarayana S, Robinson PC, Saad N, Le Cao KA, Brown MA. Diffusion-weighted Imaging Is a Sensitive and Specific Magnetic Resonance Sequence in the Diagnosis of Ankylosing Spondylitis. J Rheumatol. 2018 Jun;45(6):771-778. doi: 10.3899/jrheum.170312. Epub 2018 Feb 15. PMID 29449501
- [Background] Chung HY, Xu X, Lau VW, Ho G, Lee KL, Li PH, Tsang HH, Kwok SK, Lau CS, Wong CS. Comparing diffusion weighted imaging with clinical and blood parameters, and with short tau inversion recovery sequence in detecting spinal and sacroiliac joint inflammation in axial spondyloarthritis. Clin Exp Rheumatol. 2017 Mar-Apr;35(2):262-269. Epub 2016 Nov 13. PMID 27908306
- [Background] Chan CWS, Tsang HHL, Li PH, Lee KH, Lau CS, Wong PYS, Chung HY. Diffusion-weighted imaging versus short tau inversion recovery sequence: Usefulness in detection of active sacroiliitis and early diagnosis of axial spondyloarthritis. PLoS One. 2018 Aug 7;13(8):e0201040. doi: 10.1371/journal.pone.0201040. eCollection 2018. PMID 30086145
- [Background] Lee KH, Chung HY, Xu X, Lau VWH, Lau CS. Apparent Diffusion Coefficient as an Imaging Biomarker for Spinal Disease Activity in Axial Spondyloarthritis. Radiology. 2019 Apr;291(1):121-128. doi: 10.1148/radiol.2019180960. Epub 2019 Feb 5. PMID 30720403
- [Background] Smolen JS, Braun J, Dougados M, Emery P, Fitzgerald O, Helliwell P, Kavanaugh A, Kvien TK, Landewe R, Luger T, Mease P, Olivieri I, Reveille J, Ritchlin C, Rudwaleit M, Schoels M, Sieper J, Wit Md, Baraliakos X, Betteridge N, Burgos-Vargas R, Collantes-Estevez E, Deodhar A, Elewaut D, Gossec L, Jongkees M, Maccarone M, Redlich K, van den Bosch F, Wei JC, Winthrop K, van der Heijde D. Treating spondyloarthritis, including ankylosing spondylitis and psoriatic arthritis, to target: recommendations of an international task force. Ann Rheum Dis. 2014 Jan;73(1):6-16. doi: 10.1136/annrheumdis-2013-203419. Epub 2013 Jun 8. PMID 23749611
- [Background] Landewe R, Sieper J, Mease P, Inman RD, Lambert RG, Deodhar A, Marzo-Ortega H, Magrey M, Kiltz U, Wang X, Li M, Zhong S, Mostafa NM, Lertratanakul A, Pangan AL, Anderson JK. Efficacy and safety of continuing versus withdrawing adalimumab therapy in maintaining remission in patients with non-radiographic axial spondyloarthritis (ABILITY-3): a multicentre, randomised, double-blind study. Lancet. 2018 Jul 14;392(10142):134-144. doi: 10.1016/S0140-6736(18)31362-X. Epub 2018 Jun 29. PMID 29961640
- [Background] Gratacos J, Pontes C, Juanola X, Sanz J, Torres F, Avendano C, Vallano A, Calvo G, de Miguel E, Sanmarti R; REDES-TNF investigators. Non-inferiority of dose reduction versus standard dosing of TNF-inhibitors in axial spondyloarthritis. Arthritis Res Ther. 2019 Jan 8;21(1):11. doi: 10.1186/s13075-018-1772-z. PMID 30621746
- [Background] Zhao M, Zhang P, Fang L, Luo Z, Gu J, Lin Z. Possible predictors for relapse from etanercept discontinuation in ankylosing spondylitis patients in remission: a three years' following-up study. Clin Rheumatol. 2018 Jan;37(1):87-92. doi: 10.1007/s10067-017-3763-x. Epub 2017 Aug 7. PMID 28785857
- [Background] Yang R, Liu H, Fan M. A quick decrease of bone marrow edema in sacroiliac joint could be served as a novel marker for dose tapering of etanercept in ankylosing spondylitis patients. Medicine (Baltimore). 2019 Mar;98(11):e14620. doi: 10.1097/MD.0000000000014620. PMID 30882628
- [Background] Nefla M, Holzinger D, Berenbaum F, Jacques C. The danger from within: alarmins in arthritis. Nat Rev Rheumatol. 2016 Nov;12(11):669-683. doi: 10.1038/nrrheum.2016.162. Epub 2016 Oct 13. PMID 27733758
- [Background] Dolcino M, Tinazzi E, Pelosi A, Patuzzo G, Moretta F, Lunardi C, Puccetti A. Gene Expression Analysis before and after Treatment with Adalimumab in Patients with Ankylosing Spondylitis Identifies Molecular Pathways Associated with Response to Therapy. Genes (Basel). 2017 Apr 24;8(4):127. doi: 10.3390/genes8040127. PMID 28441778
- [Background] Almasi S, Aslani S, Poormoghim H, Jamshidi AR, Poursani S, Mahmoudi M. Gene Expression Profiling of Toll-Like Receptor 4 and 5 in Peripheral Blood Mononuclear Cells in Rheumatic Disorders: Ankylosing Spondylitis and Rheumatoid Arthritis. Iran J Allergy Asthma Immunol. 2016 Feb;15(1):87-92. No abstract available. PMID 26996117
- [Background] De Rycke L, Vandooren B, Kruithof E, De Keyser F, Veys EM, Baeten D. Tumor necrosis factor alpha blockade treatment down-modulates the increased systemic and local expression of Toll-like receptor 2 and Toll-like receptor 4 in spondylarthropathy. Arthritis Rheum. 2005 Jul;52(7):2146-58. doi: 10.1002/art.21155. PMID 15986373
- [Background] Yang ZX, Liang Y, Zhu Y, Li C, Zhang LZ, Zeng XM, Zhong RQ. Increased expression of Toll-like receptor 4 in peripheral blood leucocytes and serum levels of some cytokines in patients with ankylosing spondylitis. Clin Exp Immunol. 2007 Jul;149(1):48-55. doi: 10.1111/j.1365-2249.2007.03396.x. Epub 2007 Apr 25. PMID 17459079
- [Background] Kiyeko GW, Hatterer E, Herren S, Di Ceglie I, van Lent PL, Reith W, Kosco-Vilbois M, Ferlin W, Shang L. Spatiotemporal expression of endogenous TLR4 ligands leads to inflammation and bone erosion in mouse collagen-induced arthritis. Eur J Immunol. 2016 Nov;46(11):2629-2638. doi: 10.1002/eji.201646453. Epub 2016 Sep 6. PMID 27510283
- [Background] Sode J, Bank S, Vogel U, Andersen PS, Sorensen SB, Bojesen AB, Andersen MR, Brandslund I, Dessau RB, Hoffmann HJ, Glintborg B, Hetland ML, Locht H, Heegaard NH, Andersen V. Genetically determined high activities of the TNF-alpha, IL23/IL17, and NFkB pathways were associated with increased risk of ankylosing spondylitis. BMC Med Genet. 2018 Sep 12;19(1):165. doi: 10.1186/s12881-018-0680-z. PMID 30208882
- [Background] Schelbergen RF, Blom AB, van den Bosch MH, Sloetjes A, Abdollahi-Roodsaz S, Schreurs BW, Mort JS, Vogl T, Roth J, van den Berg WB, van Lent PL. Alarmins S100A8 and S100A9 elicit a catabolic effect in human osteoarthritic chondrocytes that is dependent on Toll-like receptor 4. Arthritis Rheum. 2012 May;64(5):1477-87. doi: 10.1002/art.33495. PMID 22127564
- [Background] Voller T, Faust A, Roth J, Schafers M, Vogl T, Hermann S. A Non-Peptidic S100A9 Specific Ligand for Optical Imaging of Phagocyte Activity In Vivo. Mol Imaging Biol. 2018 Jun;20(3):407-416. doi: 10.1007/s11307-017-1148-9. PMID 29185197
- [Background] Turina MC, Sieper J, Yeremenko N, Conrad K, Haibel H, Rudwaleit M, Baeten D, Poddubnyy D. Calprotectin serum level is an independent marker for radiographic spinal progression in axial spondyloarthritis. Ann Rheum Dis. 2014 Sep;73(9):1746-8. doi: 10.1136/annrheumdis-2014-205506. Epub 2014 May 20. No abstract available. PMID 24845387
- [Background] Hu H, Du F, Zhang S, Zhang W. Serum calprotectin correlates with risk and disease severity of ankylosing spondylitis and its change during first month might predict favorable response to treatment. Mod Rheumatol. 2019 Sep;29(5):836-842. doi: 10.1080/14397595.2018.1519103. Epub 2019 Jan 3. PMID 30175641
- [Background] Olofsson T, Lindqvist E, Mogard E, Andreasson K, Marsal J, Geijer M, Kristensen LE, Wallman JK. Elevated faecal calprotectin is linked to worse disease status in axial spondyloarthritis: results from the SPARTAKUS cohort. Rheumatology (Oxford). 2019 Jul 1;58(7):1176-1187. doi: 10.1093/rheumatology/key427. PMID 30649509
- [Background] Gupta L, Bhattacharya S, Agarwal V, Aggarwal A. Elevated levels of serum MRP8/14 in ankylosing spondylitis: associated with peripheral arthritis and active disease. Clin Rheumatol. 2016 Dec;35(12):3075-3079. doi: 10.1007/s10067-016-3448-x. Epub 2016 Oct 13. PMID 27738838
- [Background] Levitova A, Hulejova H, Spiritovic M, Pavelka K, Senolt L, Husakova M. Clinical improvement and reduction in serum calprotectin levels after an intensive exercise programme for patients with ankylosing spondylitis and non-radiographic axial spondyloarthritis. Arthritis Res Ther. 2016 Nov 25;18(1):275. doi: 10.1186/s13075-016-1180-1. PMID 27887637
- [Background] Huang J, Yin Z, Song G, Cui S, Jiang J, Zhang L. Discriminating Value of Calprotectin in Disease Activity and Progression of Nonradiographic Axial Spondyloarthritis and Ankylosing Spondylitis. Dis Markers. 2017;2017:7574147. doi: 10.1155/2017/7574147. Epub 2017 May 24. PMID 28630526
- [Background] Paramarta JE, Turina MC, Noordenbos T, Heijda TF, Blijdorp IC, Yeremenko N, Baeten D. A proof-of-concept study with the tyrosine kinase inhibitor nilotinib in spondyloarthritis. J Transl Med. 2016 Oct 27;14(1):308. doi: 10.1186/s12967-016-1050-2. PMID 27784336
- [Background] Schelbergen RF, de Munter W, van den Bosch MH, Lafeber FP, Sloetjes A, Vogl T, Roth J, van den Berg WB, van der Kraan PM, Blom AB, van Lent PL. Alarmins S100A8/S100A9 aggravate osteophyte formation in experimental osteoarthritis and predict osteophyte progression in early human symptomatic osteoarthritis. Ann Rheum Dis. 2016 Jan;75(1):218-25. doi: 10.1136/annrheumdis-2014-205480. Epub 2014 Sep 1. PMID 25180294
- [Background] Geven EJ, van den Bosch MH, Di Ceglie I, Ascone G, Abdollahi-Roodsaz S, Sloetjes AW, Hermann S, Schafers M, van de Loo FA, van der Kraan PM, Koenders MI, Foell D, Roth J, Vogl T, van Lent PL. S100A8/A9, a potent serum and molecular imaging biomarker for synovial inflammation and joint destruction in seronegative experimental arthritis. Arthritis Res Ther. 2016 Oct 24;18(1):247. doi: 10.1186/s13075-016-1121-z. PMID 27776554
- [Background] van Lent PL, Blom AB, Schelbergen RF, Sloetjes A, Lafeber FP, Lems WF, Cats H, Vogl T, Roth J, van den Berg WB. Active involvement of alarmins S100A8 and S100A9 in the regulation of synovial activation and joint destruction during mouse and human osteoarthritis. Arthritis Rheum. 2012 May;64(5):1466-76. doi: 10.1002/art.34315. PMID 22143922
- [Background] van den Bosch MH, Blom AB, Schelbergen RF, Vogl T, Roth JP, Sloetjes AW, van den Berg WB, van der Kraan PM, van Lent PL. Induction of Canonical Wnt Signaling by the Alarmins S100A8/A9 in Murine Knee Joints: Implications for Osteoarthritis. Arthritis Rheumatol. 2016 Jan;68(1):152-63. doi: 10.1002/art.39420. PMID 26360647
- [Background] Schelbergen RF, van Dalen S, ter Huurne M, Roth J, Vogl T, Noel D, Jorgensen C, van den Berg WB, van de Loo FA, Blom AB, van Lent PL. Treatment efficacy of adipose-derived stem cells in experimental osteoarthritis is driven by high synovial activation and reflected by S100A8/A9 serum levels. Osteoarthritis Cartilage. 2014 Aug;22(8):1158-66. doi: 10.1016/j.joca.2014.05.022. Epub 2014 Jun 10. PMID 24928317
- [Background] Koenders MI, Marijnissen RJ, Devesa I, Lubberts E, Joosten LA, Roth J, van Lent PL, van de Loo FA, van den Berg WB. Tumor necrosis factor-interleukin-17 interplay induces S100A8, interleukin-1beta, and matrix metalloproteinases, and drives irreversible cartilage destruction in murine arthritis: rationale for combination treatment during arthritis. Arthritis Rheum. 2011 Aug;63(8):2329-39. doi: 10.1002/art.30418. PMID 21520013
- [Background] Zhu B, Zhu Q, Li N, Wu T, Liu S, Liu S. Association of serum/plasma high mobility group box 1 with autoimmune diseases: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Jul;97(29):e11531. doi: 10.1097/MD.0000000000011531. PMID 30024540
- [Background] Chen Y, Sun W, Li S, Ni J, Su Y, Wang C, Luo X, Tu W, Shen G, Gong F, Zheng F, Dong L. Preliminary study of high mobility group box chromosomal protein 1(HMGB1) in ankylosing spondylitis patients. Clin Exp Rheumatol. 2015 Mar-Apr;33(2):187-94. Epub 2015 Jan 20. PMID 25602579
- [Background] Wang C, Miao Y, Wu X, Huang Y, Sun M, Zhu Y, Zheng F, Sun W, Dong L. Serum HMGB1 Serves as a Novel Laboratory Indicator Reflecting Disease Activity and Treatment Response in Ankylosing Spondylitis Patients. J Immunol Res. 2016;2016:6537248. doi: 10.1155/2016/6537248. Epub 2016 Oct 5. PMID 27800496
- [Background] Oktayoglu P, Em S, Tahtasiz M, Bozkurt M, Ucar D, Yazmalar L, Nas K, Yardimeden I, Cevik F, Celik Y, Mete N. Elevated serum levels of high mobility group box protein 1 (HMGB1) in patients with ankylosing spondylitis and its association with disease activity and quality of life. Rheumatol Int. 2013 May;33(5):1327-31. doi: 10.1007/s00296-012-2578-y. Epub 2012 Nov 10. PMID 23143556
- [Background] Hou C, Luan L, Ren C. Oxidized low-density lipoprotein promotes osteoclast differentiation from CD68 positive mononuclear cells by regulating HMGB1 release. Biochem Biophys Res Commun. 2018 Jan 1;495(1):1356-1362. doi: 10.1016/j.bbrc.2017.11.083. Epub 2017 Nov 14. PMID 29146189
- [Background] Hasegawa M, Yoshida T, Sudo A. Role of tenascin-C in articular cartilage. Mod Rheumatol. 2018 Mar;28(2):215-220. doi: 10.1080/14397595.2017.1349560. Epub 2017 Jul 19. PMID 28722504
- [Background] Okamura N, Hasegawa M, Nakoshi Y, Iino T, Sudo A, Imanaka-Yoshida K, Yoshida T, Uchida A. Deficiency of tenascin-C delays articular cartilage repair in mice. Osteoarthritis Cartilage. 2010 Jun;18(6):839-48. doi: 10.1016/j.joca.2009.08.013. Epub 2009 Sep 6. PMID 19747998
- [Background] Matsui Y, Hasegawa M, Iino T, Imanaka-Yoshida K, Yoshida T, Sudo A. Tenascin-C Prevents Articular Cartilage Degeneration in Murine Osteoarthritis Models. Cartilage. 2018 Jan;9(1):80-88. doi: 10.1177/1947603516681134. Epub 2016 Dec 4. PMID 29219023
- [Background] Gupta L, Bhattacharya S, Aggarwal A. Tenascin-C, a biomarker of disease activity in early ankylosing spondylitis. Clin Rheumatol. 2018 May;37(5):1401-1405. doi: 10.1007/s10067-017-3938-5. Epub 2018 Jan 8. PMID 29313272
- [Background] Midwood K, Sacre S, Piccinini AM, Inglis J, Trebaul A, Chan E, Drexler S, Sofat N, Kashiwagi M, Orend G, Brennan F, Foxwell B. Tenascin-C is an endogenous activator of Toll-like receptor 4 that is essential for maintaining inflammation in arthritic joint disease. Nat Med. 2009 Jul;15(7):774-80. doi: 10.1038/nm.1987. Epub 2009 Jun 28. PMID 19561617
- [Background] Sofat N, Robertson SD, Hermansson M, Jones J, Mitchell P, Wait R. Tenascin-C fragments are endogenous inducers of cartilage matrix degradation. Rheumatol Int. 2012 Sep;32(9):2809-17. doi: 10.1007/s00296-011-2067-8. Epub 2011 Aug 27. PMID 21874326
- [Background] Schwenzer A, Jiang X, Mikuls TR, Payne JB, Sayles HR, Quirke AM, Kessler BM, Fischer R, Venables PJ, Lundberg K, Midwood KS. Identification of an immunodominant peptide from citrullinated tenascin-C as a major target for autoantibodies in rheumatoid arthritis. Ann Rheum Dis. 2016 Oct;75(10):1876-83. doi: 10.1136/annrheumdis-2015-208495. Epub 2015 Dec 9. PMID 26659718
- [Background] Cutolo M, Soldano S, Paolino S. Potential roles for tenascin in (very) early diagnosis and treatment of rheumatoid arthritis. Ann Rheum Dis. 2020 Apr;79(4):e42. doi: 10.1136/annrheumdis-2019-215063. Epub 2019 Feb 1. No abstract available. PMID 30709814
- [Background] Maksymowych WP. Biomarkers for Diagnosis of Axial Spondyloarthritis, Disease Activity, Prognosis, and Prediction of Response to Therapy. Front Immunol. 2019 Mar 7;10:305. doi: 10.3389/fimmu.2019.00305. eCollection 2019. PMID 30899255